CLINICAL TRIAL: NCT05496998
Title: Transcatheter Mitral Valve Replacement With the Medtronic Intrepid™ TMVR Transfemoral System in Patients With Severe Symptomatic Mitral Regurgitation - APOLLO-EU Trial
Brief Title: Transcatheter Mitral Valve Replacement in Patients With Severe Symptomatic Mitral Regurgitation - APOLLO-EU Trial
Acronym: APOLLO-EU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT22008TMV005
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation
Keywords: mitral; valve; regurgitation; TMVR; Intrepid™; symptomatic; severe
MeSH Terms: conditions — Mitral Valve Insufficiency; Gastroesophageal Reflux; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Subjects with moderate-to-severe or severe symptomatic mitral regurgitation, or moderate symptomatic mitral regurgitation combined with mitral stenosis in the presence of MAC who, by agreement of the local site multidisciplinary heart team experienced in mitral valve therapies, are unsuitable for treatment with approved transcatheter repair or surgical mitral valve intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Medtronic Intrepid™ TMVR TF System (Experimental): Medtronic Intrepid™ TMVR TF System
  Interventions: Device: Medtronic Intrepid™ TMVR TF System

INTERVENTIONS:
Device: Medtronic Intrepid™ TMVR TF System — Patients with moderate-to-severe or severe symptomatic mitral regurgitation, or moderate symptomatic mitral regurgitation combined with mitral stenosis in the presence of MAC will have a Transcatheter Mitral Valve Replacement with the Medtronic Intrepid™ TMVR Transfemoral System

SUMMARY:
Evaluate the safety and efficacy of Medtronic Intrepid™ TMVR TF System in patients with moderate-to-severe or severe symptomatic mitral regurgitation, or moderate symptomatic mitral regurgitation combined with mitral stenosis in the presence of MAC who, by agreement of the local site multidisciplinary heart team experienced in mitral valve therapies, are unsuitable for treatment with approved transcatheter repair or surgical mitral valve intervention.

DETAILED DESCRIPTION:
Prospective, single-arm, multi-center, interventional, pre-market trial

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate-to-severe or severe symptomatic mitral regurgitation as defined by the American Society of Echocardiography 2017 Guidelines and Standards - Recommendations for Non-invasive Evaluation of Native Valvular Regurgitation, or subject has moderate symptomatic mitral regurgitation combined with mitral stenosis with the presence of MAC
* Local site multidisciplinary heart team experienced in mitral valve therapies agrees that patient is unsuitable for treatment with approved transcatheter repair or conventional mitral valve surgery
* Subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits
* Subject meets the legal minimum age to provide informed consent based on local regulatory requirements
* Subjects anatomically suitable for the Medtronic Intrepid™ TMVR TF System

Exclusion Criteria:

* Estimated life expectancy of less than 24 months
* Currently surgically implanted mitral valve
* Prior transcatheter mitral valve procedure with device currently implanted
* Anatomic contraindications
* Anatomically prohibitive mitral annular calcification (MAC)
* Aortic valve disease requiring intervention or previous intervention within 90 days of enrollment
* LVEF < 25% (measured by resting transthoracic echocardiogram), patients with LVEF 25 - <30% will be further evaluated by the Screening Committee for approval (Right Ventricular Dysfunction, pulmonary hypertension, and left ventricular function)
* Left ventricular end diastolic diameter (LVEDD) > 75mm
* Need for emergent or urgent surgery
* Hemodynamic instability
* History of bleeding diathesis or coagulopathy
* End stage renal disease
* Liver failure
* Frailty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Safety: all-cause mortality at 1-year post-procedure. | 1 year
  Rate of all-cause mortality at 1-year post-procedure.
Efficacy: Percentage of subjects with none/trace or mild mitral regurgitation at 30 days post-procedure. | 30 days
  Percentage of subjects with none/trace or mild mitral regurgitation at 30 days post-procedure as assessed by the Echocardiography Core Laboratory.

SECONDARY OUTCOMES:
Rate of all-cause mortality (Safety). | 30 days
  Rate of all-cause mortality at 30 days post-procedure.
Disabling stroke (Safety). | 30 days
  Rate of disabling stroke at 30 days post-procedure.
Acute Kidney Injury (stage 3 or with renal replacement) (Safety). | 30 days
  Rate of acute kidney injury (stage 3 or with renal replacement) at 30 days post-procedure.
Reoperation or reintervention (Safety). | 30 days
  Rate of reoperation or reintervention at 30 days post-procedure.
Major access site vascular complications (Safety). | 30 days
  Number of major access site vascular complications at 30 days post-procedure.
Mitral valve regurgitation (Efficacy). | 1 year
  Degree of mitral valve regurgitation at 1 year as assessed by the Echocardiography Core Laboratory.
NYHA functional class (Efficacy). | 1 year
  Change in NYHA functional class at 1 year (Efficacy).
Quality of Life (QoL) as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) (Efficacy). | 1 year
  Change of Quality of Life (QoL) at 1 year as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ). KCCQ scores are scaled from 0 to 100, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Cardiovascular hospitalizations (Efficacy). | 1 year
  Cardiovascular hospitalizations through 1 year (Efficacy).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Modine, Prof., Principal Investigator — University Hospital, Bordeaux; von Bardeleben, Prof., Principal Investigator — University Medical Center Mainz
Locations (37):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- France (8):
  - Clinique Pasteur, Toulouse, Cedex 03
  - CHU Bordeaux, Bordeaux, Pessac Cedex
  - Henri-Mondor University Hospital, Créteil
  - CHU Timone, Marseille
  - CHU de Nantes, Nantes
  - CHU Rennes - Pontchaillou Hospital, Rennes
  - Centre Cardiologique du Nord (CCN), Saint-Denis
  - CHRU de Tours, Tours
- Germany (9):
  - Heart and Diabetes Center NRW, Bad Oeynhausen
  - Deutsches Herzzentrum der Charité (DHZC), Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg
  - Herzzentrum Leipzig, Leipzig
  - University Medical Center Mainz, Mainz
  - Deutsches Herzzentrum München, München
  - LMU Clinic of University Hospital München, München
  - Universitätsklinikum Ulm, Ulm
- Italy (5):
  - Azienda Ospedaliero - Universitaria di Bologna - Policlinico S.Orsola Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - IRCCS Policlinico San Donato, San Donato Milanese
- Netherlands (3):
  - Catharina Hospital, Eindhoven
  - St. Antonius Hospital, Nieuwegein
  - Erasmus University Medical Center, Rotterdam
- Spain (4):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Central University Hospital of Asturias, Oviedo
  - University Hospital Alvaro Cunqueiro, Vigo
- Universitätsspital Bern, Bern, Switzerland
- United Kingdom (4):
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - Leeds General Infirmary, Leeds
  - Guys & St Thomas NHS Foundation Trust - St Thomas Hospital London, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang GHL, Rajagopal V, Sorajja P, Bajwa T, Gooley R, Walton A, Modine T, Ng MK, Williams MR, Zajarias A, Hildick-Smith D, Tchetche D, Spargias K, Rajani R, Bapat VN, De Backer O, Blackman D, McCarthy P, Laine M, Jain R, Martin R, Thaden JJ, Marka NA, Mack M, Adams DH, Leon MB, Reardon MJ. Five-year outcomes of the early-generation Intrepid transapical transcatheter mitral valve replacement system. EuroIntervention. 2026 Feb 2;22(3):e172-e182. doi: 10.4244/EIJ-D-25-01133. PMID 41251714